CLINICAL TRIAL: NCT01052740
Title: X-Ray Mammography Standard of Care Protocol
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100042; 10-CC-0042
Record Dates: First submitted 2010-01-16; First posted 2010-01-20 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-09-20

CONDITIONS: Breast Cancer; Invasive Carcinoma; In Situ Carcinoma; Fibrocystic Changes; Atypical Ductal Hyperplasia
Keywords: Breast Cancer; Mammography; Screening
MeSH Terms: conditions — Breast Neoplasms; Carcinoma in Situ; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* X-ray mammography is the standard method for breast cancer screening. It is a noninvasive test using x-rays to take pictures of breast tissue and detect any abnormalities.
* The National Institutes of Health (NIH) Clinical Center has a breast imaging unit that has been accredited by the American College of Radiology. To maintain accreditation, the unit must recruit a certain number of women to have clinical mammograms each year in order to maintain a high level of clinical skills and experience for the radiologists and technologists.

Objectives:

- To create a state-of-the-art mammography unit at the NIH Clinical Center in order to maintain American College of Radiology accreditation of the NIH breast imaging facility.

Eligibility:

- Women who are eligible for breast cancer screening because of family cancer history, genetic test results, or previous instances of cancer. Participants may not be pregnant or nursing at the time of the screening.

Design:

* Participants will provide a brief medical history on arrival at the NIH breast imaging unit.
* Each participant will have a standard mammogram performed by a radiology technician.
* If the study is normal, participants will be told that no further evaluation will be performed. If the results indicate a need for further imaging or tissue biopsy, participants may elect to return to the care of their primary physician or to receive further follow-up at the NIH Clinical Center.

DETAILED DESCRIPTION:
Background:

A mammography facility in the Clinical Center of the National Institutes of Health (NIH) is present in order to facilitate breast cancer research programs. The American College of Radiology mammography accreditation program (1992 mammography Quality Standards Act (MQSA) (1-3)) has established national standards for site accreditation for mammography. A key requirement is to perform a minimum number of mammography examinations in the facility per year. Minimum examination volumes are required to maintain expertise of the facility staff for maintaining facility accreditation and compliance with Food and Drug Administration (FDA) requirements.

Objectives:

Our primary aim is a protocol to maintain accreditation of the NIH breast imaging facility in the Clinical Center of NIH.

Eligibility:

Women who are clinically indicated for screening mammography according to the National Comprehensive Cancer Network (NCCN) guidelines (3) and the American Cancer Society guidelines.

Design:

A standard of care protocol to perform standard clinically indicated mammography exams. We are expected to recruit 1000 patient /year.

ELIGIBILITY:
* INCLUSION CRITERIA:

Women who are clinically indicated for screening mammography according to the National Comprehensive Cancer Network (NCCN) guidelines (3) and the American Cancer Society guidelines:

1. All women who fall under the ACS mammography guidelines
2. Women younger than 40 years but with more than 20% lifetime risk for developing breast cancer:

   1. Prior personal history of prior thoracic radiation therapy between the age of 10 and 30, such as for Hodgkin's disease. In this case, women are eligible beginning 8-10 years after radiotherapy or at age 40, whichever comes first.
   2. 5-year risk of invasive breast cancer (greater than or equal to 1.7% of women greater than or equal to 35 years or women who have a life time risk greater than 20% as defined by models that are largely dependent on family history.
   3. Strong family history;

   i. First degree relative diagnosed with breast, ovarian, fallopian tube, or primary peritoneal cancer.

   ii. Individual from families known to have BRCA 1 or 2 gene mutation.

   iii. Close male blood relative with breast cancer.

   d. Genetic predisposition;

   i. Carry or have first-degree relative who carries a genetic mutation in the BRCA 1 or 2 genes.

   ii. Carry or have a first-degree relative who carries a genetic mutation in the TP53 or PTEN genes (Li-Fraumeni syndrome and Cowden Bannayan-Riley-Ruvalcaba syndromes).

   e. A personal history of Lobular carcinoma in situ (LCIS) and/or atypical ductal hyperplasia (ADH)

   f. Prior personal history of breast cancer or ovarian cancer.

   i. Starting at the age of 25 year for Hereditary breast and ovarian cancer patients.

   ii. 5-10 years prior to youngest breast cancer case for strong family history or other genetic predisposition.

   g. Woman and Minorities

   EXCLUSION CRITERIA:

   Pregnant or lactating subjects.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2009-12-30; Study Completion 2011-09-20

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Destouet JM, Bassett LW, Yaffe MJ, Butler PF, Wilcox PA. The ACR's Mammography Accreditation Program: ten years of experience since MQSA. J Am Coll Radiol. 2005 Jul;2(7):585-94. doi: 10.1016/j.jacr.2004.12.005. PMID 17411883
- [Background] Geller BM, Ichikawa LE, Buist DS, Sickles EA, Carney PA, Yankaskas BC, Dignan M, Kerlikowske K, Yabroff KR, Barlow W, Rosenberg RD; Breast Cancer Surveillance Consortium. Improving the concordance of mammography assessment and management recommendations. Radiology. 2006 Oct;241(1):67-75. doi: 10.1148/radiol.2411051375. PMID 16990672
- [Background] Belkacemi Y, Bousquet G, Marsiglia H, Ray-Coquard I, Magne N, Malard Y, Lacroix M, Gutierrez C, Senkus E, Christie D, Drumea K, Lagneau E, Kadish SP, Scandolaro L, Azria D, Ozsahin M. Phyllodes tumor of the breast. Int J Radiat Oncol Biol Phys. 2008 Feb 1;70(2):492-500. doi: 10.1016/j.ijrobp.2007.06.059. Epub 2007 Oct 10. PMID 17931796